CLINICAL TRIAL: NCT05257499
Title: In-person Versus Online Debriefing in the Simulation Sessions of the Helping Babies Breathe Course: A Randomized Controlled Trial
Brief Title: In-person Versus Online Debriefing in HBB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Lama Charafeddine, Associate Professor of Clinical Pediatrics and Neonatology, Director of the Neonatal Resuscitation Education Program, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SBS-2021-0193
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2022-02

CONDITIONS: Neonatal Respiratory Distress
Keywords: Online debriefing; In person debriefing; Helping babies breathe; Debriefing; Simulation training
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- On line debfriefing (Experimental): Participants in this group will practice the skills taught as above but in the presence of the same certified instructor who will guide them throughout all the steps of HBB using a virtual platform (Webex® or Zoom®).
  Interventions: Behavioral: On line debriefing
- In person debriefing (No Intervention): Participants in this group will practice the skills taught in the virtual class on the neonatal mannequin. They are expected to work as a small group of 3 to 4 at a time. They will receive coaching, debriefing and feedback from a certified instructor who will conduct the traditional in-person training with face-to-face feedback and debriefing.

INTERVENTIONS:
Behavioral: On line debriefing — Online Debriefing in the Simulation Sessions of the Helping Babies Breathe Course
  Arms: On line debfriefing

SUMMARY:
The objective of this study is to assess the effectiveness of online formative feedback and debriefing on nursing and medical students enrolled in the HBB course in comparison to traditional face-to-face feedback. The working hypothesis is that online feedback and debriefing during hands-on training sessions are as effective as face-to-face feedback and debriefing in teaching clinical skills to medical and nursing students.

DETAILED DESCRIPTION:
Online learning has become an integral part of education, especially during the ongoing COVID19 pandemic that has imposed a limit on live interactions. This observation holds true in the medical education system which uses the flipped classroom model to teach essential practical skills. Studies have shown that this model is associated with improved learning and student satisfaction. In such a model, debriefing and feedback comprise a main part of the teaching process, and these interactions are usually conducted in person. One helpful skill offered to nursing and medical students is Helping Babies Breathe (HBB), which is an evidence-based educational program training first-line birth attendants to initiate effective resuscitation of a newborn in the first minute of life. The investigators propose to incorporate online feedback as part of the HBB course at the American University of Beirut. In this non-inferiority randomized controlled trial, the investigators will study the effectiveness of online formative feedback and debriefing on nursing and medical students enrolled in the HBB course in comparison to traditional face-to-face feedback. The working hypothesis is that internet-based live feedback and debriefing are as effective as face-to-face interactions when teaching clinical skills to nursing and medical students. This work will aid in developing a reliable online curriculum that can be extrapolated to other courses and institutions, thus broadening the reach of medical education in the times of physical distancing.

ELIGIBILITY:
Inclusion Criteria:

* Nurses and medical students

Exclusion Criteria:

* Attended resuscitation course

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Objective Structured Clinical Examination (OSCE) score | One month
  The OSCE of all participants will be videotaped without showing any identifier. Grading of the OSCE will be done by an independent instructor blinded to group assignments.
  OSCE is graded over 100. Grades equal of higher than 80% are considered for passing.

SECONDARY OUTCOMES:
Student satisfaction | One month
  A questionnaire accompanied with a standardized Debriefing Assessment for Simulation in Healthcare Student Version will be used.

CONTACTS AND LOCATIONS:
Locations (2):
- Lebanon (2):
  - American University of Beirut, Beirut, Beyrouth
  - American University of Beirut, Beirut, Hamra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Odongkara B, Tylleskar T, Pejovic N, Achora V, Mukunya D, Ndeezi G, Tumwine JK, Nankabirwa V. Adding video-debriefing to Helping-Babies-Breathe training enhanced retention of neonatal resuscitation knowledge and skills among health workers in Uganda: a cluster randomized trial. Glob Health Action. 2020 Dec 31;13(1):1743496. doi: 10.1080/16549716.2020.1743496. PMID 32524895
- [Background] Sait MS, Siddiqui Z, Ashraf Y. Advances in medical education and practice: student perceptions of the flipped classroom. Adv Med Educ Pract. 2017 May 2;8:317-320. doi: 10.2147/AMEP.S133328. eCollection 2017. No abstract available. PMID 28496377
- [Background] Mehta NB, Hull AL, Young JB, Stoller JK. Just imagine: new paradigms for medical education. Acad Med. 2013 Oct;88(10):1418-23. doi: 10.1097/ACM.0b013e3182a36a07. PMID 23969368
- [Derived] Kfoury P, Maalouf F, Nasser F, Gulgulian T, Charafeddine L. In-Person Versus Online Training in Simulations of Helping Babies Breathe: A Randomized Controlled Trial. Cureus. 2024 Jul 16;16(7):e64677. doi: 10.7759/cureus.64677. eCollection 2024 Jul. PMID 39149645